CLINICAL TRIAL: NCT01312857
Title: A Randomized Phase II Study of Hepatic Arterial Infusion With Intravenous Irinotecan, 5FU and Leucovorin With or Without Panitumumab, in Patients With Wild Type RAS Who Have Resected Hepatic Metastases From Colorectal Cancer
Brief Title: Study of Hepatic Arterial Infusion With Intravenous Irinotecan, 5FU and Leucovorin With or Without Panitumumab, in Patients With Wild Type RAS Who Have Resected Hepatic Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-137
Record Dates: First submitted 2011-03-08; First posted 2011-03-11 (Estimated); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colon; rectal; liver; AMG 954 (Panitumumab); DEXAMETHASONE; FLOXURIDINE; FLUOROURACIL; IRINOTECAN (CPT-11) CAMPTOSAR; LEUCOVORIN; 10-137
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

ARMS (2):
- Randomization to panitumumab (Experimental): Patients whose liver metastases have been completely resected will be randomized Arm A will receive Panitumumab in addition to HAI FUDR/Dexamethasone plus systemic CPT-11/5FU/LV
  Interventions: Drug: panitumumab
- Randomization to No Panitumumab (Experimental): Patients whose liver metastases have been completely resected will be randomized and patients randomized to Arm B will receive HAI FUDR/Dex plus systemic CPT-11/5FU/LV alone.
  Interventions: Drug: Randomization to No Panitumumab

INTERVENTIONS:
Drug: panitumumab — All patients receive HAI FUDR (0.12 mg/kg/day X kg X pump volume) / pump flow rate and Dexamethasone flat dose of 25 mg on days 1.
  All patients receive CPT-11 (150 mg/m2 IV over 30 min to an hour), Leucovorin (400 mg/m2 IV, over 30 min to an hour) and 5FU (1000 mg/m2/day continuous infusion over two days) on days 15 and 29 Randomization to panitumumab 6 mg/kg day 15 and 29 Each cycle repeats every 36 days for a total of 6 cycles
  Arms: Randomization to panitumumab
Drug: Randomization to No Panitumumab — All patients receive HAI FUDR (0.12 mg/kg/day X kg X pump volume) / pump flow rate and Dexamethasone flat dose of 25 mg on days 1.
  All patients receive CPT-11 (150 mg/m2 IV over 30 min to an hour), Leucovorin (400 mg/m2 IV, over 30 min to an hour) and 5FU (1000 mg/m2/day continuous infusion over two days) on days 15 and 29 Randomization (to no panitumumab) Each cycle repeats every 36 days for a total of 6 cycles
  Arms: Randomization to No Panitumumab

SUMMARY:
The purpose of this study is to see if Panitumumab plus the other treatments will increase the time of remission. Remission means that there is no sign of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed colorectal adenocarcinoma metastatic to the liver with no clinical or radiographic evidence of extrahepatic disease. Confirmation of diagnosis must be performed at MSKCC.
* Completely resected hepatic metastases without current evidence of other metastatic disease.
* Lab values ≤ 14 days prior to treatment start:
* WBC ≥ 3.0 K/uL
* ANC > 1.5 K/uL
* Platelets ≥ 100,000/uL
* Creatinine <1.5 mg/dL
* HGB ≥ 9 gm/dL Renal function (≤ 14 days prior to treatment start).
* Creatinine ≤1.5 mg/dL or creatinine clearance ≥ 50 mL/min calculated by the

Cockcroft-Gault method as follows:

* Male creatinine clearance = (140 -age in years) x (weight in Kg) / (serum Cr in mg/dl x 72)
* Female creatinine clearance = (140 - age in years) x (weight in Kg) x 0.85 / (serum Cr in mg/dl x 72) (use of creatinine clearance per protocol based on chemotherapy regimen) Hepatic function, as follows: (≤ 14 days prior to treatment start)
* Aspartate aminotransferase (AST) (≤ 5 x ULN)
* Alanine aminotransferase (ALT) (≤ 5 x ULN)
* Total Bilirubin ≤ 1.5 mg/dl
* Magnesium ≥ lower limit of normal (≤ 48 hours prior to treatment start.)
* Calcium ≥ lower limit of normal (≤ 48 hours prior to treatment start.)
* Prior chemotherapy is acceptable if last dose given ≥ 3 weeks prior to registration to this study. [Note: no chemotherapy to be given after resection of liver lesions prior to treatment on this study.]
* Any investigational agent is acceptable if administered ≤ 30 days before registration
* KPS ≥ 60% (ECOG (or Karnofsky) performance status (preferably 0 or 1/≥ 60% for Karnofsky)
* Histologically confirmed all RAS wild type.
* Paraffin-embedded tumor tissue obtained from the primary tumor or metastasis (Prior to

Exclusion Criteria:

* Patients < 18 years of age.
* Prior radiation to the liver (Prior radiation therapy to the pelvis is acceptable if completed at least 4 weeks prior to registration.)
* Active infection, ascites, hepatic encephalopathy.
* Prior treatment with HAI FUDR.
* Patients who have had prior anti EGFR antibody therapy inhibitors and who have not responded to this treatment will be excluded. However, patients who have responded to prior anti-EGFR therapy are eligible.)
* Female patients who are pregnant or lactating - or planning to become pregnant within 6 months after the end of the treatment (female patients of child-bearing potential must have negative pregnancy test ≤ 72 hours before registration).
* If a patient has any serious medical problems which may preclude receiving this type of treatment.
* Patients with current evidence of hepatitis A, B, C (ie, active hepatitis)
* Patients with history or known presence of primary CNS tumors, seizures not well controlled with standard medical therapy, or history of stroke will also be excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Panitumumab.
* Serious or non-healing active wound, ulcer, or bone fracture.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* Patients who have a diagnosis of Gilbert's disease.
* History of other malignancy, except:
* Malignancy treated with curative intent and with no known active disease present for ≥ 3 years prior to registration and felt to be at low risk for recurrence by the treating physician
* Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease
* Adequately treated cervical carcinoma in situ without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-03-07 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kemeny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Kemeny NE, Chou JF, Capanu M, Chatila WK, Shi H, Sanchez-Vega F, Kingham TP, Connell LC, Jarnagin WR, D'Angelica MI. A Randomized Phase II Trial of Adjuvant Hepatic Arterial Infusion and Systemic Therapy With or Without Panitumumab After Hepatic Resection of KRAS Wild-type Colorectal Cancer. Ann Surg. 2021 Aug 1;274(2):248-254. doi: 10.1097/SLA.0000000000004923. PMID 33938493
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomization to Panitumumab: Patients whose liver metastases have been completely resected will be randomized Arm A will receive Panitumumab in addition to HAI FUDR/Dexamethasone plus systemic CPT-11/5FU/LV
  panitumumab: All patients receive HAI FUDR (0.12 mg/kg/day X kg X pump volume) / pump flow rate and Dexamethasone flat dose of 25 mg on days 1.
  All patients receive CPT-11 (150 mg/m2 IV over 30 min to an hour), Leucovorin (400 mg/m2 IV, over 30 min to an hour) and 5FU (1000 mg/m2/day continuous infusion over two days) on days 15 and 29 Randomization to panitumumab 6 mg/kg day 15 and 29 Each cycle repeats every 36 days for a total of 6 cycles
- Randomization to No Panitumumab: Patients whose liver metastases have been completely resected will be randomized and patients randomized to Arm B will receive HAI FUDR/Dex plus systemic CPT-11/5FU/LV alone.
  Randomization to No Panitumumab: All patients receive HAI FUDR (0.12 mg/kg/day X kg X pump volume) / pump flow rate and Dexamethasone flat dose of 25 mg on days 1.
  All patients receive CPT-11 (150 mg/m2 IV over 30 min to an hour), Leucovorin (400 mg/m2 IV, over 30 min to an hour) and 5FU (1000 mg/m2/day continuous infusion over two days) on days 15 and 29 Randomization (to no panitumumab) Each cycle repeats every 36 days for a total of 6 cycles
Period: Overall Study
Arm/Group | Randomization to Panitumumab | Randomization to No Panitumumab
Started | 37 | 38
Completed | 29 | 37
Not Completed | 8 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomization to Panitumumab | Randomization to No Panitumumab | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Median (Full Range); unit: years] | 52 [27 to 75] | 53 [33 to 75] | 53 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 25 | 21 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 34 | 34 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 6 | 6
  White | 34 | 27 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Participants With Recurrence Free Survival for Colorectal Cancer Participants With Resected Liver Metastases
Description: to determine if panitumumab with Hepatic Arterial Infusion (HAI) in combination with systemic chemotherapy can increase the recurrence free survival (RFS) for colorectal cancer patients with resected liver metastases
Time Frame: 15 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomization to Panitumumab | Randomization to No Panitumumab
Number analyzed (Participants) | 37 | 38
percentage of participants | 69 [53 to 82] | 47 [32 to 63]

2. Secondary Outcome: Number of Participants Evaluated for Toxicity as Per the NCI Common Toxicity Criteria
Description: Toxicities will be recorded as adverse events on the Adverse Event case report form and must be graded using The National Cancer Institute's Common Toxicity Criteria (CTC)version 4.0 with the exception of skin- or nail-related toxicities, which must be graded using CTC version 3.0 with modifications
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization to Panitumumab | Randomization to No Panitumumab
Number analyzed (Participants) | 37 | 38
Participants | 37 | 38

3. Secondary Outcome: Participant Survival
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization to Panitumumab | Randomization to No Panitumumab
Number analyzed (Participants) | 37 | 38
Participants
  Alive | 22 | 11
  Dead | 15 | 27

4. Secondary Outcome: Number of Participants With Tumor Tissue Expression of Predictive Makers
Description: (such as NRAS, BRAF, PIK3CA, AKT1 and MEK1), and correlate with patient progression and survival following therapy.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization to Panitumumab | Randomization to No Panitumumab
Number analyzed (Participants) | 37 | 38
Participants
  NRAS | 1 | 1
  BRAF | 0 | 2
  PIK3CA | 3 | 8
  AKT1 | 0 | 0
  MEK1 | 0 | 0
  Participants without predictive tumor markers | 33 | 27

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Randomization to Panitumumab | Randomization to No Panitumumab
All-Cause Mortality (participants affected / at risk) | 15/37 | 27/38
Serious Adverse Events (participants affected / at risk) | 14/37 | 6/38
Other Adverse Events (participants affected / at risk) | 27/37 | 26/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization to Panitumumab (N=37) | Randomization to No Panitumumab (N=38)
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hyperbilirubinemia (Investigations) | 1 | 0
Chills (General disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Fever (General disorders) | 3 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Leukocytes (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Pain - Other (General disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 3
Thromboembolic event (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Weight loss (Investigations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization to Panitumumab (N=37) | Randomization to No Panitumumab (N=38)
Alanine aminotransferase increased (Investigations) | 12 | 11
Alkaline phosphatase increased (Investigations) | 4 | 3
Blood bilirubin increased (Investigations) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 8 | 4
Rash (Skin and subcutaneous tissue disorders) | 9 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Lymphopenia (Investigations) | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0
Paronychia (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT01312857/Prot_SAP_000.pdf